CLINICAL TRIAL: NCT01141569
Title: A Phase 2 Study of RO4929097 (IND 109291) in Patients With Advanced Renal Cell Carcinoma (RCC, NOS 10038415) That Has Progressed After VEGF/VEGFR Directed Therapy
Brief Title: A Study of RO4929097 in Patients With Advanced Renal Cell Carcinoma That Have Failed Vascular Endothelial Growth Factor (VEGF)/Vascular Endothelial Growth Factor Receptor (VEGFR) Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03068; NCI-2012-03068 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHL-077 (Other: University Health Network-Princess Margaret Hospital); 8563 (Other: CTEP); N01CM00032 (NIH); NCT01145521 (obsolete NCT alias)
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (1):
- Treatment (RO4929097) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: RO4929097
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
The purpose of this study is to evaluate the activity of RO4929097 in renal cell carcinoma patients that have failed therapy with VEGF/VEGFR directed agents.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the objective response rate of RO4929097 in patients with advanced kidney cancer and failure of anti-VEGF directed therapy.

SECONDARY OBJECTIVES:

I. To assess the antitumor activity of RO4929097 through secondary endpoints including: duration of radiologic response, rate of disease stabilizations, rate of tumor control rate (CR+PR+SD), and progression-free & overall survival rates.

II. To assess the safety and tolerability of single agent RO4929097 in patients with advanced RCC.

III. To explore expression of Notch biomarkers in RCC patients and their potential interaction with RO4929097 response and toxicity.

OUTLINE:

Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 orally (PO) on days 1-3, 8-10, and 15-17. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed predominant clear cell, renal cell carcinoma, NOS, that is recurrent or metastatic
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan; scans must be completed within 4 weeks prior to starting study treatment
* Patients must have had one prior therapy for non-resectable renal cell carcinoma with a VEGF/VEGFR targeted therapy (e.g. sunitinib, sorafenib, other VEGFR tyrosine kinase inhibitor, or bevacizumab)

  * Prior treatment with mTOR inhibitors (Everolimus, Temsirolimus, or rapamycin) for non-resectable disease is permitted
  * Prior immunotherapy is permitted
  * Only one line of prior VEGF/VEGFR is permitted
* Life expectancy of greater than 3 months
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Patients must have normal organ and marrow function as defined below (within 7days prior to starting study treatment):
* Hemoglobin >= 90 g/L
* Absolute granulocyte count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.25 x ULN
* AST (SGOT)/ALT (SGPT) =< 1.5 x institutional upper limit of normal (=< 5 x ULN for patients with liver metastases)
* Creatinine =< within institutional normal limits OR creatinine clearance >= mL/min/1.73 m^2 for patients with creatinine levels above institutional (using Cockcroft-Gault formula)
* Patients must have no serious medical conditions such as myocardial infarction within 6 months prior to entry, congestive heart failure, unstable angina, active cardiomyopathy, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, psychiatric illness, or any other medical conditions that might be aggravated by treatment or limit compliance
* Patients must have no active malignancy at any other site
* Patients must be able to take oral medication and have no evidence of bowel obstruction
* The effects of RO4929097 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because Notch signal pathway inhibitors are known to be teratogenic, if women of childbearing potential do not abstain from sexual activity (documentation that they have been abstinent from sexual activity at least 4 weeks prior to study entry) they must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry; women of childbearing potential be can either be abstinent or use two forms of contraception for the duration of study participation, and be either abstinent or use two forms of contraception for at least 12 months post-treatment; men must use condoms when sexually active with women for the duration of study participation and at least 12 months post-treatment

  * Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately
  * Pregnancy Testing; women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of RO4929097; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097, the investigator or clinical staff must confirm and document the patient's use of two contraceptive methods or abstinence, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097
  * Female patients of childbearing potential are defined as follows:

    * Patients with regular menses
    * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
    * Women who have had tubal ligation
  * Female patients may be considered to NOT be of childbearing potential for the following reasons:

    * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
    * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive months
    * Pre-pubertal females; the parent or guardian of young female patients who have not yet started menstruation should verify that menstruation has not begun; if a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients must not have had major surgery, chemotherapy, or radiation therapy within 4 weeks of starting the study treatment (6 weeks for nitrosoureas or mitomycin C); prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that had not been irradiated; patients must have recovered from the toxic effects from any prior therapy to =< grade 1, except alopecia
* Patients may not be receiving any other investigational agents concurrently
* Patients with controlled brain metastases (no radiographic progression following radiation and/or surgical treatment and no neurological signs or symptoms) that are clinically and radiologically stable for at least 6 months will be allowed but must NOT be currently taking corticosteroids (e.g. dexamethasone) to control neurologic symptoms of brain metastases

  * Patients with unstable or symptomatic brain metastases, spinal core compression, or carcinomatosis meningitis, or evidence of brain or leptomeningeal disease on screening CT or MRI scan are excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or other agents used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* Preclinical studies indicate that RO4929097 is a substrate of CYP3A4 and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Patients who are serologically positive for Hepatitis A, B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because RO4929097 is a Notch pathway-inhibiting agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with RO4929097, breastfeeding should be discontinued if the mother is treated with RO4929097; these potential risks may also apply to other agents used in this study
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with RO4929097; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Cardiovascular: baseline (within 7days prior to starting study treatment) QTc > 450 msec (male) or QTc > 470 msec (female)

  * History of risk factors for QT interval prolongation, including, but not limited to family or personal history of long QT syndrome, recurrent syncope without known etiology or sudden unexpected death
  * History of Torsades de Pointes or other significant cardiac arrhythmias or the need for concomitant meds with known potential to prolong QT interval or antiarrhythmics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Kollmannsberger, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (4):
- Canada (4):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute-General Division, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (RO4929097)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 60 [49 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  Canada | 12

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (PR + CR) Using RECIST
Description: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: Up to 12 months
Population: Patients that had PR or CR (Objective response)
Measure: Number; unit: participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 12
participants | 0

2. Secondary Outcome: Time to Progression
Description: Time to Progression is duration of time from start of treatment to time of progression
Time Frame: Up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 12
months | 1.2 [0.8 to 2.6]

3. Secondary Outcome: Frequency and Severity of Adverse Events
Description: Tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.
Time Frame: Up to 12 months
Population: Number analyzed is number of participants who experienced the adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 12
Participants
  Fatigue: Grade 1-2 | 12
  Fatigue: Grade 3-4 | 0
  Insomnia: number analyzed (Participants) | 10
  Insomnia: Grade 1-2 | 10
  Insomnia: Grade 3-4 | 0
  Anorexia: number analyzed (Participants) | 9
  Anorexia: Grade 1-2 | 9
  Anorexia: Grade 3-4 | 0
  Anemia: number analyzed (Participants) | 8
  Anemia: Grade 1-2 | 8
  Anemia: Grade 3-4 | 0
  Nausea: number analyzed (Participants) | 7
  Nausea: Grade 1-2 | 7
  Nausea: Grade 3-4 | 0
  Creatinine increased: number analyzed (Participants) | 6
  Creatinine increased: Grade 1-2 | 6
  Creatinine increased: Grade 3-4 | 0
  Pruritis: number analyzed (Participants) | 6
  Pruritis: Grade 1-2 | 6
  Pruritis: Grade 3-4 | 0
  Lymphocyte count decreased: number analyzed (Participants) | 9
  Lymphocyte count decreased: Grade 1-2 | 7
  Lymphocyte count decreased: Grade 3-4 | 2
  Hypoalbuminemia: number analyzed (Participants) | 6
  Hypoalbuminemia: Grade 1-2 | 6
  Hypoalbuminemia: Grade 3-4 | 0
  Edema limbs: number analyzed (Participants) | 5
  Edema limbs: Grade 1-2 | 5
  Edema limbs: Grade 3-4 | 0
  Hyponatremia: number analyzed (Participants) | 6
  Hyponatremia: Grade 1-2 | 4
  Hyponatremia: Grade 3-4 | 2
  Hypophosphatemia: number analyzed (Participants) | 4
  Hypophosphatemia: Grade 1-2 | 3
  Hypophosphatemia: Grade 3-4 | 1
  Dyspnea: number analyzed (Participants) | 5
  Dyspnea: Grade 1-2 | 5
  Dyspnea: Grade 3-4 | 0
  Bone Pain: number analyzed (Participants) | 6
  Bone Pain: Grade 1-2 | 4
  Bone Pain: Grade 3-4 | 2
  AST increased: number analyzed (Participants) | 5
  AST increased: Grade 1-2 | 5
  AST increased: Grade 3-4 | 0
  ALP Increased: number analyzed (Participants) | 5
  ALP Increased: Grade 1-2 | 5
  ALP Increased: Grade 3-4 | 0
  Hypertension: number analyzed (Participants) | 5
  Hypertension: Grade 1-2 | 3
  Hypertension: Grade 3-4 | 2
  Flank Pain: number analyzed (Participants) | 4
  Flank Pain: Grade 1-2 | 4
  Flank Pain: Grade 3-4 | 0
  Vomiting: number analyzed (Participants) | 4
  Vomiting: Grade 1-2 | 4
  Vomiting: Grade 3-4 | 0
  ALT increased: number analyzed (Participants) | 4
  ALT increased: Grade 1-2 | 4
  ALT increased: Grade 3-4 | 0

4. Secondary Outcome: Progression-free Survival Rate
Description: Progression-free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: From start of treatment to time of progression or death, whichever occurs first, assessed up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 12
months | 1.2 [0.8 to 2.6]

5. Secondary Outcome: Rate of Disease Stabilizations
Description: Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: Up to 12 months
Population: Number of patients who had Stable disease
Measure: Number; unit: participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 12
participants | 4

6. Secondary Outcome: Tumor Control Rate (CR + PR + SD)
Description: Tumor control rate is defined as the sum of objective response rate (CR+PR) and stable disease (SD) rate.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097)
Number analyzed (Participants) | 12
Participants | 4

ADVERSE EVENTS:
Arm/Group | Treatment (RO4929097)
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (RO4929097) (N=12)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (RO4929097) (N=12)
Fatigue (General disorders) | 12 (12)
Insomnia (Psychiatric disorders) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 7 (7)
Creatinine increased (Investigations) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6)
Lymphocyte count decreased (Investigations) | 9 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (6)
Edema limbs (General disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
AST increased (Investigations) | 5 (5)
ALP increased (Investigations) | 5 (5)
Hypertension (Vascular disorders) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Vomiting (General disorders) | 4 (4)
ALT increased (Investigations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less